CLINICAL TRIAL: NCT06474429
Title: Assessing the Functional Movement Screen as a Reliable Physical Therapy Discharge Criteria for Chronic Lower Back Pain Patients
Status: Recruiting | Type: Observational
Sponsor: Texas Back Institute (Other)
Responsible Party: Sponsor
Other Study IDs: 2169799
Record Dates: First submitted 2024-06-19; First posted 2024-06-25 (Actual); Last update posted 2024-06-25 (Actual); Status verified 2024-03

CONDITIONS: Chronic Lower Back Pain
Keywords: Chronic Lower Back Pain; Physical Therapy; Discharge

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- CLBP Patients: Patients who have experienced LBP for longer than three months and are undergoing physical therapy for their symptoms will be recruited from the Texas Back Institute.

SUMMARY:
Overview of Research Design and Objectives

This study is a prospective, concurrent cohort study aimed at evaluating the reliability of the Functional Movement Screen (FMS) as a discharge criterion for patients with chronic lower back pain (LBP) undergoing physical therapy. The primary objective is to identify a benchmark FMS score that correlates with a low risk of recurrence and high levels of functional performance post-discharge.

Specific Aims and Hypotheses

The study specifically aims to:

Assess the effectiveness of FMS in determining discharge readiness for chronic LBP patients.

The hypothesis is that a specific threshold score on the FMS can reliably indicate a patient's readiness for discharge, reducing the risk of recurrence and ensuring better long-term functional outcomes.

Rationale for the Study

Chronic LBP is a prevalent condition requiring multidisciplinary management. The FMS, widely used in athletic and military settings, has potential utility in clinical management of chronic LBP, particularly in establishing discharge criteria. This study seeks to explore this potential, addressing a gap in evidence regarding discharge benchmarks for chronic LBP patients.

Procedures

The study involves 50 chronic LBP patients from the Texas Back Institute. Participants will undergo their standard physical therapy regimen, supplemented by regular FMS assessments to evaluate discharge readiness. Assessments include a series of functional tasks, with scores ranging from 0 to 3 for each task, culminating in a total possible score of 21.

Risks and Anticipated Benefits

Risks are minimal, akin to those in low-intensity exercises. Benefits include improved discharge criteria for chronic LBP patients, potentially enhancing long-term outcomes. All procedures adhere to Good Clinical Practice and Health Insurance Portability and Accountability Act guidelines. This study's risks include potential loss of confidentiality, psychological, and physical risks. Physical risks are minimal, similar to those in low-intensity exercises like squatting and lunging. To protect confidentiality, data will be managed in compliance with Good Clinical Practice and HIPAA guidelines, with encryption and secure storage. Psychological and physical risks are mitigated through thorough instruction, practice trials, and breaks for participants. Additionally, trained study personnel can terminate a participant's involvement at any point for safety reasons.

Outcomes

The study will report on the average FMS score correlating with discharge readiness and the variance in scores across different functional assessments.

Statistical Analysis

Data will be analyzed using descriptive statistics, correlation analysis, and repeated measures ANOVA or Friedman Test, with a significance level set at α=0.05.

Completion Time

The study is expected to complete enrollment within two years.

Abbreviations and Terms

LBP: Lower Back Pain FMS: Functional Movement Screen PROM: Patient-Reported Outcome Measures VAS: Visual Analog Scale ODI: Oswestry Disability Index ANOVA: Analysis of Variance PROMIS: Patient-Reported Outcomes Measurement Information System®

ELIGIBILITY:
* Non-surgical patients who have had lower back pain for >3 months
* Patients who include and are between the ages of 18 and 49
* Patients with a BMI of <30
* Not pregnant with no plans of becoming pregnant during the duration of the study
* Be able and willing to understand and sign consent for study participation
* Be physically able to comply with study protocol requirements
* Not have had recent surgeries or have confounding factors that would keep them from being able to perform any portion of the FMS assessment

Ages: 18 Years to 49 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Patients who have experienced LBP for longer than three months and are undergoing physical therapy for their symptoms will be recruited from the Texas Back Institute.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2024-04-26 (Actual); Primary Completion 2026-03-08 (Estimated); Study Completion 2026-09-08 (Estimated)

PRIMARY OUTCOMES:
Average FMS Scores | From enrollment to the end of treatment at 12 weeks
  e study will report on the average FMS score correlating with discharge readiness and the variance in scores across different functional assessments.

CONTACTS AND LOCATIONS:
Overall Officials: Steven Kight, PT, Principal Investigator — Texas Back Institute
Locations (1):
- Texas Back Institute, Plano, Texas, United States

IPD SHARING:
Plan to Share IPD: Undecided